CLINICAL TRIAL: NCT03229096
Title: Apatinib Plus XELOX Regime as Neoadjuvant Therapy in Locally Advanced Gastric Cancer Patients With Lymph Node Metastasis
Brief Title: Apatinib Plus XELOX as Neoadjuvant Therapy in Locally Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSGC-002
Record Dates: First submitted 2017-07-22; First posted 2017-07-25 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Chemotherapy Effect; Chemotherapeutic Toxicity; Gastric Cancer
Keywords: gastric cancer; neoadjuvant chemotherapy; apatinib
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib; XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib plus XELOX (Experimental): Patients will be given the perioperative chemotherapy of Apatinib plus XELOX once recruited
  Interventions: Drug: Apatinib plus XELOX

INTERVENTIONS:
Drug: Apatinib plus XELOX — three weeks is one cycle, 4 cycles followed by radical gastrectomy. Apatinib: 250 mg, p.o., qd, every 3 weeks for the first two cycles. if no level 3 or severer AEs happened, change apatinib to 500mg, p.o.,qd, otherwise keep 250mg in the third cycle. no apatinib in the fourth cycle.
  Capecitabine: 1000mg/m2, p.o., bid, D1-14, every 3 weeks (treatment for 2 weeks and rest 1 week).
  Oxaliplatin: 130mg/m2, i.v. over 2h, D1, every 3 weeks.

SUMMARY:
Apatinib plus XELOX regime as Neoadjuvant Therapy in Locally Advanced Gastric Cancer PatientsWith lymph node metastasis

DETAILED DESCRIPTION:
This is a Single-center, Open-label, Single-arm,Non-randomized exploratory clinical trial evaluating the efficacy and safety of Apatinib plus XELOX regime as Neoadjuvant Therapy in Locally Advanced Gastric Cancer Patients With lymph node metastasis

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, age ≥18 years.
2. Karnofsky score 70%.
3. Histologically confirmed adenocarcinoma of gastric cancer with Lauren classification Clinically diagnosed stage T2-T4aN+M0 according to CT/MRI scan.
4. At least one measurable and evaluable disease based on response evaluation criteria in solid tumors (RECIST v1.1), that is one or more perigastric lymph note were greater than or equal to 1.5cm in diameter.
5. Laparoscopic exploration confirms no peritoneal metastasis and negative peritoneal lavage.
6. Physical condition and adequate organ function to ensure the success of abdominal surgery.
7. Adequate hematological function: Neutrophil count ≥ 1.5 × 109/L, Platelets ≥ 100 × 109/L and Hemoglobin ≥8g/dL. Adequate liver function: Total bilirubin ≤ 1.5 × upper limit of normal (ULN); AST (SGOT) and ALT (SGPT) < 2.5 × ULN. ALP ≤ 2.5 × upper limit of normal (ULN); ALB ≥30g/L.Adequate renal function: Serum creatinine ≤ 1 x ULN, and serum albumin≥30g/L.
8. Life expectancy of more than 5 years without serious concomitant diseases.
9. Written (signed) informed consent.
10. Able to comply with study and follow-up procedures.
11. Consent to provide tissue sample.

Exclusion Criteria:

1. Pregnant or lactating women.
2. pregnancy tests before entering the group (in serum) of the childbearing age women were positive, or no pregnancy tests.
3. patients with distant metastases or local unresectable factors.
4. tumor stage considered as cT1 by imaging or ultrasound gastroscopy.
5. Patients who received prior anti-tumor therapy including cytotoxic chemotherapy, radiotherapy, hormonal therapy and immunotherapy.
6. History of other malignancies within the last 5 years except cured basal cell carcinoma of skin and carcinoma in situ of uterine cervix.
7. History of significant neurological or mental disorder, including seizures or dementia, which may interfere compliance and sign of consent inform.
8. Unstable, persistent cardiac disease despite medicinal treatment; myocardial infarction within 12 months before the start of the trial.
9. Patients with poor-controlled arterial hypertension (systolic pressure ≥ 140 mmHg and/or diastolic pressure ≥ 90 mm Hg) despite standard medical management.
10. Ileus, chronic inflammatory intestinal disease or extensive resection of the small intestine and other disorders which limit drug absorption.
11. Patients who experienced GI bleeding within two weeks, or with high risk of bleeding.
12. Patients with symptomatic peripheral neuropathy NCI CTC version> 1.0 grade, except only the deficiency of Deep tendon reflex.
13. Organ transplant patient need immunosuppression treatment.
14. Active or uncontrolled severe infection or other severe and /or uncontrolled diseases
15. Patients with moderate or severe chronic kidney disease estimated glomerular filtration rate≤50 ml/min or serum creatinine ≥the upper limit of normal(ULN),
16. deficiency of dihydropyrimidine dehydrogenase (DPD)
17. Allergy to the drugs in this protocol
18. Less than 4 weeks from the last clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 3 months
  Both CR and PR according to Response Evaluation Criteria in Solid Tumors RECIST Version 1.1

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 30 days
  The safety of the the perioperative treatment, percentage of grade 3 or 4 adverse events as safety profile of perioperative treatments
Pathological response rate (pRR) | 30 days
  Briefly, pathCR (Pathological complete rate) was defined as an absence of carcinoma cells in the primary site, and pathologic partial response (pathPR) was defined as less than 10% residual carcinoma cells in the specimen.
3-year disease free survival rate | 3 years
3-year overall survival rate | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- ZhongShan hospital FuDan university, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Sasako M, Sano T, Yamamoto S, Kurokawa Y, Nashimoto A, Kurita A, Hiratsuka M, Tsujinaka T, Kinoshita T, Arai K, Yamamura Y, Okajima K; Japan Clinical Oncology Group. D2 lymphadenectomy alone or with para-aortic nodal dissection for gastric cancer. N Engl J Med. 2008 Jul 31;359(5):453-62. doi: 10.1056/NEJMoa0707035. PMID 18669424
- [Background] Songun I, Putter H, Kranenbarg EM, Sasako M, van de Velde CJ. Surgical treatment of gastric cancer: 15-year follow-up results of the randomised nationwide Dutch D1D2 trial. Lancet Oncol. 2010 May;11(5):439-49. doi: 10.1016/S1470-2045(10)70070-X. Epub 2010 Apr 19. PMID 20409751
- [Background] Fujitani K, Yang HK, Mizusawa J, Kim YW, Terashima M, Han SU, Iwasaki Y, Hyung WJ, Takagane A, Park DJ, Yoshikawa T, Hahn S, Nakamura K, Park CH, Kurokawa Y, Bang YJ, Park BJ, Sasako M, Tsujinaka T; REGATTA study investigators. Gastrectomy plus chemotherapy versus chemotherapy alone for advanced gastric cancer with a single non-curable factor (REGATTA): a phase 3, randomised controlled trial. Lancet Oncol. 2016 Mar;17(3):309-318. doi: 10.1016/S1470-2045(15)00553-7. Epub 2016 Jan 26. PMID 26822397
- [Background] Sano T, Coit DG, Kim HH, Roviello F, Kassab P, Wittekind C, Yamamoto Y, Ohashi Y. Proposal of a new stage grouping of gastric cancer for TNM classification: International Gastric Cancer Association staging project. Gastric Cancer. 2017 Mar;20(2):217-225. doi: 10.1007/s10120-016-0601-9. Epub 2016 Feb 20. PMID 26897166
- [Background] Yoshikawa T, Sasako M, Yamamoto S, Sano T, Imamura H, Fujitani K, Oshita H, Ito S, Kawashima Y, Fukushima N. Phase II study of neoadjuvant chemotherapy and extended surgery for locally advanced gastric cancer. Br J Surg. 2009 Sep;96(9):1015-22. doi: 10.1002/bjs.6665. PMID 19644974
- [Background] Cunningham D, Allum WH, Stenning SP, Thompson JN, Van de Velde CJ, Nicolson M, Scarffe JH, Lofts FJ, Falk SJ, Iveson TJ, Smith DB, Langley RE, Verma M, Weeden S, Chua YJ, MAGIC Trial Participants. Perioperative chemotherapy versus surgery alone for resectable gastroesophageal cancer. N Engl J Med. 2006 Jul 6;355(1):11-20. doi: 10.1056/NEJMoa055531. PMID 16822992
- [Background] Iwasaki Y, Sasako M, Yamamoto S, Nakamura K, Sano T, Katai H, Tsujinaka T, Nashimoto A, Fukushima N, Tsuburaya A; Gastric Cancer Surgical Study Group of Japan Clinical Oncology Group. Phase II study of preoperative chemotherapy with S-1 and cisplatin followed by gastrectomy for clinically resectable type 4 and large type 3 gastric cancers (JCOG0210). J Surg Oncol. 2013 Jun;107(7):741-5. doi: 10.1002/jso.23301. Epub 2013 Feb 11. PMID 23400787
- [Background] Inoue K, Nakane Y, Kogire M, Fujitani K, Kimura Y, Imamura H, Tamura S, Okano S, Kwon AH, Kurokawa Y, Shimokawa T, Takiuchi H, Tsujinaka T, Furukawa H. Phase II trial of preoperative S-1 plus cisplatin followed by surgery for initially unresectable locally advanced gastric cancer. Eur J Surg Oncol. 2012 Feb;38(2):143-9. doi: 10.1016/j.ejso.2011.11.009. Epub 2011 Dec 9. PMID 22154885
- [Background] Koizumi W, Narahara H, Hara T, Takagane A, Akiya T, Takagi M, Miyashita K, Nishizaki T, Kobayashi O, Takiyama W, Toh Y, Nagaie T, Takagi S, Yamamura Y, Yanaoka K, Orita H, Takeuchi M. S-1 plus cisplatin versus S-1 alone for first-line treatment of advanced gastric cancer (SPIRITS trial): a phase III trial. Lancet Oncol. 2008 Mar;9(3):215-21. doi: 10.1016/S1470-2045(08)70035-4. Epub 2008 Feb 20. PMID 18282805
- [Background] Boku N, Yamamoto S, Fukuda H, Shirao K, Doi T, Sawaki A, Koizumi W, Saito H, Yamaguchi K, Takiuchi H, Nasu J, Ohtsu A; Gastrointestinal Oncology Study Group of the Japan Clinical Oncology Group. Fluorouracil versus combination of irinotecan plus cisplatin versus S-1 in metastatic gastric cancer: a randomised phase 3 study. Lancet Oncol. 2009 Nov;10(11):1063-9. doi: 10.1016/S1470-2045(09)70259-1. Epub 2009 Oct 7. PMID 19818685
- [Background] Tsuburaya A, Mizusawa J, Tanaka Y, Fukushima N, Nashimoto A, Sasako M; Stomach Cancer Study Group of the Japan Clinical Oncology Group. Neoadjuvant chemotherapy with S-1 and cisplatin followed by D2 gastrectomy with para-aortic lymph node dissection for gastric cancer with extensive lymph node metastasis. Br J Surg. 2014 May;101(6):653-60. doi: 10.1002/bjs.9484. Epub 2014 Mar 25. PMID 24668391
- [Background] Ito S, Sano T, Mizusawa J, Takahari D, Katayama H, Katai H, Kawashima Y, Kinoshita T, Terashima M, Nashimoto A, Nakamori M, Onaya H, Sasako M. A phase II study of preoperative chemotherapy with docetaxel, cisplatin, and S-1 followed by gastrectomy with D2 plus para-aortic lymph node dissection for gastric cancer with extensive lymph node metastasis: JCOG1002. Gastric Cancer. 2017 Mar;20(2):322-331. doi: 10.1007/s10120-016-0619-z. Epub 2016 Jun 14. PMID 27299887
- [Background] Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A, Lordick F, Ohtsu A, Omuro Y, Satoh T, Aprile G, Kulikov E, Hill J, Lehle M, Ruschoff J, Kang YK; ToGA Trial Investigators. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet. 2010 Aug 28;376(9742):687-97. doi: 10.1016/S0140-6736(10)61121-X. Epub 2010 Aug 19. PMID 20728210
- [Background] Wilke H, Muro K, Van Cutsem E, Oh SC, Bodoky G, Shimada Y, Hironaka S, Sugimoto N, Lipatov O, Kim TY, Cunningham D, Rougier P, Komatsu Y, Ajani J, Emig M, Carlesi R, Ferry D, Chandrawansa K, Schwartz JD, Ohtsu A; RAINBOW Study Group. Ramucirumab plus paclitaxel versus placebo plus paclitaxel in patients with previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (RAINBOW): a double-blind, randomised phase 3 trial. Lancet Oncol. 2014 Oct;15(11):1224-35. doi: 10.1016/S1470-2045(14)70420-6. Epub 2014 Sep 17. PMID 25240821
- [Background] Li J, Qin S, Xu J, Xiong J, Wu C, Bai Y, Liu W, Tong J, Liu Y, Xu R, Wang Z, Wang Q, Ouyang X, Yang Y, Ba Y, Liang J, Lin X, Luo D, Zheng R, Wang X, Sun G, Wang L, Zheng L, Guo H, Wu J, Xu N, Yang J, Zhang H, Cheng Y, Wang N, Chen L, Fan Z, Sun P, Yu H. Randomized, Double-Blind, Placebo-Controlled Phase III Trial of Apatinib in Patients With Chemotherapy-Refractory Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction. J Clin Oncol. 2016 May 1;34(13):1448-54. doi: 10.1200/JCO.2015.63.5995. Epub 2016 Feb 16. PMID 26884585
- [Background] Okines AF, Langley RE, Thompson LC, Stenning SP, Stevenson L, Falk S, Seymour M, Coxon F, Middleton GW, Smith D, Evans L, Slater S, Waters J, Ford D, Hall M, Iveson TJ, Petty RD, Plummer C, Allum WH, Blazeby JM, Griffin M, Cunningham D. Bevacizumab with peri-operative epirubicin, cisplatin and capecitabine (ECX) in localised gastro-oesophageal adenocarcinoma: a safety report. Ann Oncol. 2013 Mar;24(3):702-9. doi: 10.1093/annonc/mds533. Epub 2012 Oct 28. PMID 23108952
- [Background] Kataoka K, Tokunaga M, Mizusawa J, Machida N, Katayama H, Shitara K, Tomita T, Nakamura K, Boku N, Sano T, Terashima M, Sasako M; Stomach Cancer Study Group/Japan Clinical Oncology Group. A randomized Phase II trial of systemic chemotherapy with and without trastuzumab followed by surgery in HER2-positive advanced gastric or esophagogastric junction adenocarcinoma with extensive lymph node metastasis: Japan Clinical Oncology Group study JCOG1301 (Trigger Study). Jpn J Clin Oncol. 2015 Nov;45(11):1082-6. doi: 10.1093/jjco/hyv134. Epub 2015 Sep 9. PMID 26355164
- [Derived] Tang Z, Wang Y, Yu Y, Cui Y, Liang L, Xu C, Shen Z, Shen K, Wang X, Liu T, Sun Y. Neoadjuvant apatinib combined with oxaliplatin and capecitabine in patients with locally advanced adenocarcinoma of stomach or gastroesophageal junction: a single-arm, open-label, phase 2 trial. BMC Med. 2022 Apr 6;20(1):107. doi: 10.1186/s12916-022-02309-0. PMID 35382819